CLINICAL TRIAL: NCT01863940
Title: Continuous Infusion of Local Anesthetic for Post-operative Pain Control in Ukraine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Political unrest in study country
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gennadiy Fuzaylov, Gennadiy Fuzaylov, M.D., Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012P002299
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wound catheter (Experimental): Wound catheters will be placed subcutaneously in the skin graft donor site in the lateral thigh while the patient remain intra-operative. The patients will receive a continuous infusion of procaine 0.5% at 4-5mL/hr using an elastomeric infusion device for 48 hours. Patients will be asked to asses pain on a 0-10 scale immediately prior to dressing changes, during dressing changes and 1 hour post dressing changes.
  Interventions: Device: Wound Catheter
- Control (No Intervention): Patients will receive the standard of care pain medication regimen of Analgin/Metamizole 1 g IM and Ketorolac 3%- 30 mg IM for post-operative pain treatment. The patients will be asked to rate pain on a scale of 0-10 immediately prior to dressing changes, during dressing changes and 1 hour after dressing changes.

INTERVENTIONS:
Device: Wound Catheter — Wound catheter placement in split thickness skin graft donor site on the thigh with continuous infusion of procaine 0.5% at 4-5cc/hr for 48 hours.
  Arms: Wound catheter

SUMMARY:
Ukraine is a newly sovereign country in Eastern Europe with a large burn population. With the collapse of the Soviet Union, burn programs have become decentralized and resources for maintaining facilities have dwindled. Patients frequently present with debilitating burn injuries and often do not receive necessary treatment secondary to limited resources and cost of treatment.

The investigators have established an annual medical mission, outreach clinic and telemedicine relationship with hospitals and burn centers in Ukraine in an effort to improve burn care. One focus is post-operative pain control. The investigators have noticed a pattern of anxiety with children from the Ukraine surrounding dressing changes which they believe this is secondary to inadequate pain control in the immediate post-operative period including the initial dressing changes.

The goal is to provide wound catheters with a continuous infusion of procaine in an attempt to reduce the pain experienced in the early post-operative period and specifically with dressing changes.

There will be 200 participants, 12-65 years old who are receiving reconstructive plastic procedure with split-thickness skin grafts from lateral thigh in the study. 100 will receive the standard pain management Analgin/Metamizole 1 g IM; Ketorolac 3%- 30 mg IM regimen and 100 will receive wound catheters with continuous procaine infusion for 48 hours with the standard Analgin/Metamizole 1 g IM; Ketorolac 3%- 30 mg IM available for breakthrough pain. Pain scores will be assessed prior to dressing change, during dressing changes and at 30 minutes and 1 hour after dressing change.

DETAILED DESCRIPTION:
There will be 200 participants, ages 12-65 years old who are receiving reconstructive plastic surgery with split-thickness skin grafts from the lateral thigh at 1 hospital in Ukrain. The first 100 will receive the standard pain regimen Analgin/Metamizole 1 g IM; Ketorolac 3%- 30 mg IM and the following 100 will receive catheters with continuous procaine infusion for 48 hours with the standard pain regimen available for breakthrough pain. All participants must be expected to remain inpatient for 48 hours post-operatively.

Participants receiving continuous infusion of local anesthetic via a wound catheter will have the ON-Q PainBuster Post-Op Pain Relief System (I-Flow Corporation) tunneled subcutaneously while the patient is intra-operative. Catheter insertion sites will be covered with Steri-strips and covered with a transparent dressing to facilitate inspection of the insertion site for any erythema or discharge. Catheters will have a 10mL procaine 0.5% bolus intra-operative followed by an infusion delivered at 4-5mL/hr delivered by an elastomeric pump. Historically patients' pain complaints arise from skin graft donor sites rather then recipient sites.

Patients will be assessed for pain scores on a scale of 0-10 (0= no pain and 10= worst possible pain) prior to dressing changes, during and 1 hour after dressing changes.

ELIGIBILITY:
Inclusion Criteria:

* those admitted for reconstructive surgery required split-thickness skin grafts from the lateral thigh as part of their management

Exclusion Criteria:

* age less than 12 years
* known allergy to local anesthetics
* pseudocholinesterase deficiency,
* documented history of dementia/psychosis/delirium
* known neurologic conditions impairing pain sensation pathways
* pregnant, and breast feeding woman due to Ukrainian requirements

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-08; Primary Completion 2022-02 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Pain Score with dressing changes | 1 hour with dressing changes over 48 hours
  Patients will be asked to record a pain score prior to dressing changes, during dressing changes and 1 hour after dressing changes for a total of 48 hours until the wound catheter is removed

CONTACTS AND LOCATIONS:
Overall Officials: Gennadiy Fuzaylov, M.D., Principal Investigator — Massachusetts General Hospital; Cheryl Bline, M.D., Study Director — Massachusetts General Hospital
Locations (1):
- Burn Unit, Municipal Hospital #8, Lviv, Ukraine

REFERENCES:
- [Background] Fuzaylov G, Driscoll DN, Volfson I. A plan to improve pediatric burn care in Ukraine. J Burn Care Res. 2013 Mar-Apr;34(2):e119-20. doi: 10.1097/BCR.0b013e318267c942. No abstract available. PMID 23202873
- [Background] Hernandez JL, Savetamal A, Crombie RE, Cholewczynski W, Atweh N, Possenti P, Schulz JT 3rd. Use of continuous local anesthetic infusion in the management of postoperative split-thickness skin graft donor site pain. J Burn Care Res. 2013 Jul-Aug;34(4):e257-62. doi: 10.1097/BCR.0b013e3182721735. PMID 23271060
- [Background] Thomas DF, Lambert WG, Williams KL. The direct perfusion of surgical wounds with local anaesthetic solution: an approach to postoperative pain? Ann R Coll Surg Engl. 1983 Jul;65(4):226-9. PMID 6347012
- [Background] Baig MK, Zmora O, Derdemezi J, Weiss EG, Nogueras JJ, Wexner SD. Use of the ON-Q pain management system is associated with decreased postoperative analgesic requirement: double blind randomized placebo pilot study. J Am Coll Surg. 2006 Feb;202(2):297-305. doi: 10.1016/j.jamcollsurg.2005.10.022. PMID 16427556
- See also: Related Info — http://www.dctohc.org